CLINICAL TRIAL: NCT05914298
Title: Analysis of the Relationship Among Height, Ulnar Length and Forearm Function in Patients With Multiple Hereditary Exostoses and Association With the Genotypic Pattern
Brief Title: Height, Ulnar Length and Forearm Function in Multiple Hereditary Exostoses
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 0012479
Record Dates: First submitted 2018-01-16; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Exostoses, Multiple Hereditary
Keywords: Multiple Hereditary Exostoses, forearm, height, ulnar length
MeSH Terms: conditions — Exostoses, Multiple Hereditary | interventions — Blood Specimen Collection; Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — blood or buccal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HME group: 204 children and adult patients with HME, admitted to our Hospital for diagnosis and treatment.
  the patients will be stratified by age in four subgroups:
  * subgroup I (0-7 Years)
  * subgroup II (8-12 Years)
  * subgroup III (13-18 Years)
  * subgroup IV (>18 Years)
  Interventions: Diagnostic Test: blood and buccal swab genetic test; Diagnostic Test: PUL; Diagnostic Test: Range of motion
- healty control group: 204 children and adult voluntary healty controls will be stratified in the same manner and matched with the population in study in order to assess normal and pathologic growth.
  Interventions: Diagnostic Test: PUL; Diagnostic Test: Range of motion

INTERVENTIONS:
Diagnostic Test: blood and buccal swab genetic test — blood samples and buccal swabs will be obtained from patients with HME in order to analyze the genotype (EXT1 or EXT2 mutations) and correlate the genotypic pattern with the phenotypic presentation
  Groups: HME group
Diagnostic Test: PUL — measurement of ulnar length with anthropometer and patient's height
Diagnostic Test: Range of motion — measurement of range of motion of elbow, forearm and wrist

SUMMARY:
the purpose of the present registry is to describe the epidemiology of forearm deformities in patients with Hereditary Multiple Exostoses and to identify, independent predictors of severity of the disease and potential association with genotypic patterns

DETAILED DESCRIPTION:
Hereditary Multiple Exostoses (HME) is a rare pediatric autosomal dominant disorder caused by loss-of-function mutations in the genes encoding the heparan sulfate (HS)-synthesizing enzymes EXT1 or EXT2. HME affects 1 in 50,000 people and has 100% penetrance but great variability in phenotypic expression. HME is characterized by formation of cartilaginous outgrowths, called osteochondromas or exostoses, next to the growth plates of many axial and appendicular skeletal elements, causing multiple, painful disfiguring and disabling skeletal deformities, and potential malignant transformation into peripherral chondrosarcoma.

The involvement of upper-limb bones by HME is associated with greater loss of function than elsewhere in the body, but even here the loss of function may be limited. Moreover, the constant relationship between height and ulnar length has long been recognized in forensic medicine and has been recently analyzed also in HME, in order to predict the clinical and functional outcomes of the upper limb.

the present registry aims to collect demographic, clinical, functional and radiographic information from patients with HME in order to establish phenotypic predictors of severity of the disease and potential association with genotypic patterns

ELIGIBILITY:
Inclusion Criteria:

- patients with HME (> 2 exostoses)

Exclusion Criteria:

* Patients with solitary exostoses
* Patients, adults or minors, who are unable to give their timely informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults Patients with HME.
Sampling Method: Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
proportional ulnar length (PUL) | 1 year
  proportional ulnar length (PUL) is the ratio between ulnar lenght and the height of the patient

SECONDARY OUTCOMES:
genotype | 1 year
  identify potential association among the genotypic pattern (EXT1 or EXT2) and phenotypic presentation
forearm function | 1 year
  elbow, forearm and wrist range of motion (ROM) measured by a goneometer
EuroQol 5D | 1 year
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol Group

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luigi Di Gennaro, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Manila Boarini, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pedrini E, De Luca A, Valente EM, Maini V, Capponcelli S, Mordenti M, Mingarelli R, Sangiorgi L, Dallapiccola B. Novel EXT1 and EXT2 mutations identified by DHPLC in Italian patients with multiple osteochondromas. Hum Mutat. 2005 Sep;26(3):280. doi: 10.1002/humu.9359. PMID 16088908
- [Result] Mordenti M, Ferrari E, Pedrini E, Fabbri N, Campanacci L, Muselli M, Sangiorgi L. Validation of a new multiple osteochondromas classification through Switching Neural Networks. Am J Med Genet A. 2013 Mar;161A(3):556-60. doi: 10.1002/ajmg.a.35819. Epub 2013 Feb 8. PMID 23401177
- [Result] Pedrini E, Jennes I, Tremosini M, Milanesi A, Mordenti M, Parra A, Sgariglia F, Zuntini M, Campanacci L, Fabbri N, Pignotti E, Wuyts W, Sangiorgi L. Genotype-phenotype correlation study in 529 patients with multiple hereditary exostoses: identification of "protective" and "risk" factors. J Bone Joint Surg Am. 2011 Dec 21;93(24):2294-302. doi: 10.2106/JBJS.J.00949. PMID 22258776
- [Result] Clement ND, Porter DE. Forearm deformity in patients with hereditary multiple exostoses: factors associated with range of motion and radial head dislocation. J Bone Joint Surg Am. 2013 Sep 4;95(17):1586-92. doi: 10.2106/JBJS.L.00736. PMID 24005199